CLINICAL TRIAL: NCT05177393
Title: Treatment Outcomes of Esophageal Cancer
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Westat (Other); African Esophageal Cancer Consortium (AfrECC) (Unknown); National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TOEC-AfrECC; 21455 (Other: University of California, San Francisco); 184510 (Other: University of California, San Francisco); 214520 (Other: University of California, San Francisco); 204510 (Other: University of California, San Francisco); 184515 (Other: University of California, San Francisco); 3P30CA082103-21SA (NIH)
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Cancer
Keywords: Treatment outcomes; Quality of life; Comparative effectiveness; Palliation
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Esophageal Cancer: Participants with esophageal cancer will be administered questionnaires, and medical charts will be accessed to collect study related data.
  Interventions: Other: Assessment of patient-reported outcomes (PROs)

INTERVENTIONS:
Other: Assessment of patient-reported outcomes (PROs) — Questionnaires will be administered to participants
  Other Names: PROs

SUMMARY:
This study will be a carried out through a prospective observational cohort design in conjunction with researchers in the African Esophageal Cancer Consortium (AfrECC). The purpose of this research is to prospectively evaluate outcomes related to existing treatment strategies for esophageal cancer (EC) at participating sites within AfrECC.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

Aim 1: To describe the types of treatments administered for all patients diagnosed with EC at participating AfrECC sites, including chemotherapeutic regimens, radiation therapy, chemo-radiotherapy, esophageal stenting, esophagectomy, and basic supportive care.

Aim 2: To evaluate the effect of different EC treatment modalities on patient reported outcomes during and after completion of treatment.

Aim 3: To measure the effect of different treatment modalities on overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histopathologically confirmed or presumptive clinical diagnosis of EC. For patients who do not have histopathologically confirmed disease, presumptive clinical diagnosis may be based upon barium swallow or endoscopy without biopsy.
* Age 18 years of age or older;

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with esophageal cancer based on histological confirmation or presumptive clinical diagnosis who reside in Kenya, Tanzania, and Malawi.
Sampling Method: Probability Sample
Enrollment: 2476 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of esophageal cancer (EC) participants receiving treatment with varying treatment modalities at participating AfrECC sites | Up to 4 years
  Descriptive statistics will be used to describe the proportion of EC patients receiving treatment with each modality at participating AfrECC sites. The investigators will assess the associations between demographic and clinicopathologic characteristic and treatment modalities employed (chemotherapy, radiotherapy, chemo-radiation, esophageal stenting, esophagectomy, supportive care alone, or a combination of these treatments)
Change in scores of the Modified Rosenblatt Index over time | Up to 4 years
  The 6-item Modified Rosenblatt Index by Rosenblatt, et al. adapted for use within a resource-limited context evaluates EC related parameters scored on a Likert scale assessing presence and severity of symptoms: Odynophagia (0=no pain on swallowing to 3=severe pain); Dysphagia (0=normal, no dysphagia to 4=unable to swallow saliva); Regurgitation (0=never to 3=constant); Chest and/or Back Pain (0=no pain to 2=pain not relieved by non-narcotics or requiring opiate medication); World Health Organization (WHO) performance status/Overall Well-Being (0="A lot better" to 4="A lot worse"). Scores will be assessed at the following time points: Baseline, 1 month and 3 months after initiation of treatment, and every 3 months thereafter.
Median Overall Survival | Up to 4 years
  Survival will be defined as the time elapsed from date of diagnosis (either confirmed or date of diagnostic modality leading to presumptive clinical diagnosis) to date of death. For participants who are not deceased, censorship will be performed on the date when the participant was last known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Buckle, MD, MPH, Principal Investigator — University of California, San Francisco; Katherine Van Loon, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (6):
- Kenya (2):
  - Tenwek Hospital, Bomet
  - Moi Teaching and Referral Hospital, Eldoret
- Kamuzu Central Hospital, Lilongwe, Malawi
- Tanzania (3):
  - Muhimbili National Hospital, Dar es Salaam
  - Ocean Road Cancer Institute, Dar es Salaam
  - Kilimanjaro Christian Medical Centre, Moshi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mulima G, Mody GN, Kaimila B, Salima A, Williams B, Paciorek A, Zhang L, Charles A, Westmoreland KD, Van Loon K, Buckle GC. Treatment Outcomes of Esophageal Cancer in Malawi: An Analysis of Overall Survival and Patient-Reported Outcomes. JCO Glob Oncol. 2025 Nov;11:e2500221. doi: 10.1200/GO-25-00221. Epub 2025 Nov 13. PMID 41232057
- [Derived] Buckle GC, Mrema A, Mwachiro M, Ringo Y, Selekwa M, Mulima G, Some FF, Mmbaga BT, Mody GN, Zhang L, Paciorek A, Akoko L, Ayuo P, Burgert S, Bukusi E, Charles A, Chepkemoi W, Chesumbai G, Kaimila B, Kenseko A, Kibwana KS, Koech D, Macharia C, Moirana EN, Mushi BP, Mremi A, Mwaiselage J, Mwanga A, Ndumbalo J, Nvakunga G, Ngoma M, Oduor M, Oloo M, Opakas J, Parker R, Seno S, Salima A, Servent F, Wandera A, Westmoreland KD, White RE, Williams B, Mmbaga EJ, Van Loon K; of the African Esophageal Cancer Consortium (AfrECC). Treatment outcomes of esophageal cancer in Eastern Africa: protocol of a multi-center, prospective, observational, open cohort study. BMC Cancer. 2022 Jan 19;22(1):82. doi: 10.1186/s12885-021-09124-5. PMID 35045815